CLINICAL TRIAL: NCT00970762
Title: Comparative Study of Org 9426 With Vecuronium Bromide (Phase III)
Brief Title: Comparative Study of Rocuronium With Vecuronium (Study 71101)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05975; 71101
Record Dates: First submitted 2009-07-23; First posted 2009-09-02 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Rocuronium; Maintenance; Vecuronium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Rocuronium 0.6 INT, 0.1 MNT (Experimental): Participants in this group received a 0.6 mg/kg intubating dose of rocuronium followed by 0.1 mg/kg maintenance dose of rocuronium.
  Interventions: Drug: Rocuronium 0.6 mg/kg intubating dose; Drug: Rocuronium 0.1 mg/kg maintenance dose
- Rocuronium 0.6 INT, 0.15 MNT (Experimental): Participants in this group received a 0.6 mg/kg intubating dose of rocuronium followed by 0.15 mg/kg maintenance dose of rocuronium.
  Interventions: Drug: Rocuronium 0.6 mg/kg intubating dose; Drug: Rocuronium 0.15 mg/kg maintenance dose
- Rocuronium 0.6 INT, 0.2 MNT (Experimental): Participants in this group received a 0.6 mg/kg intubating dose of rocuronium followed by 0.2 mg/kg maintenance dose of rocuronium.
  Interventions: Drug: Rocuronium 0.6 mg/kg intubating dose; Drug: Rocuronium 0.2 mg/kg maintenance
- Rocuronium 0.9 INT, 0.1 MNT (Experimental): Participants in this group received a 0.9 mg/kg intubating dose of rocuronium followed by 0.1 mg/kg maintenance dose of rocuronium.
  Interventions: Drug: Rocuronium 0.9 mg/kg intubating dose; Drug: Rocuronium 0.1 mg/kg maintenance dose
- Rocuronium 0.9 INT, 0.15 MNT (Experimental): Participants in this group received a 0.9 mg/kg intubating dose of rocuronium followed by 0.15 mg/kg maintenance dose of rocuronium.
  Interventions: Drug: Rocuronium 0.9 mg/kg intubating dose; Drug: Rocuronium 0.15 mg/kg maintenance dose
- Rocuronium 0.9 INT, 0.2 MNT (Experimental): Participants in this group received a 0.9 mg/kg intubating dose of rocuronium followed by 0.2 mg/kg maintenance dose of rocuronium.
  Interventions: Drug: Rocuronium 0.9 mg/kg intubating dose; Drug: Rocuronium 0.2 mg/kg maintenance
- Vecuronium 0.1 INT, 0.025 MNT (Active Comparator): Participants in this group received a 0.1 mg/kg intubating dose of vecuronium followed by 0.025 mg/kg maintenance dose of vecuronium.
  Interventions: Drug: Vecuronium 0.1 mg/kg intubating dose; Drug: Vecuronium 0.025 mg/kg maintenance dose

INTERVENTIONS:
Drug: Rocuronium 0.6 mg/kg intubating dose — Rocuronium 0.6 mg/kg intubating dose
  Other Names: Zemuron; Org 9426
  Arms: Rocuronium 0.6 INT, 0.1 MNT; Rocuronium 0.6 INT, 0.15 MNT; Rocuronium 0.6 INT, 0.2 MNT
Drug: Rocuronium 0.9 mg/kg intubating dose — 0.9 mg/kg intubating dose of rocuronium
  Other Names: Zemuron; Org 9426
  Arms: Rocuronium 0.9 INT, 0.1 MNT; Rocuronium 0.9 INT, 0.15 MNT; Rocuronium 0.9 INT, 0.2 MNT
Drug: Rocuronium 0.1 mg/kg maintenance dose — Rocuronium 0.1 mg/kg maintenance dose following the intubating dose.
  Other Names: Zemuron; Org 9426
  Arms: Rocuronium 0.6 INT, 0.1 MNT; Rocuronium 0.9 INT, 0.1 MNT
Drug: Rocuronium 0.15 mg/kg maintenance dose — Rocuronium 0.15 mg/kg maintenance dose following the intubating dose
  Other Names: Zemuron; Org 9426
  Arms: Rocuronium 0.6 INT, 0.15 MNT; Rocuronium 0.9 INT, 0.15 MNT
Drug: Rocuronium 0.2 mg/kg maintenance — Rocuronium 0.2 mg/kg maintenance dose following the intubating dose
  Other Names: Zemuron; Org 9426
  Arms: Rocuronium 0.6 INT, 0.2 MNT; Rocuronium 0.9 INT, 0.2 MNT
Drug: Vecuronium 0.1 mg/kg intubating dose — Vecuronium 0.1 mg/kg intubating dose
  Other Names: Norcuron
  Arms: Vecuronium 0.1 INT, 0.025 MNT
Drug: Vecuronium 0.025 mg/kg maintenance dose — Vecuronium 0.025 mg/kg maintenance dose following the intubating dose
  Other Names: Norcuron
  Arms: Vecuronium 0.1 INT, 0.025 MNT

SUMMARY:
This study was conducted to determine and compare the safety and effectiveness of two neuromuscular blockers (rocuronium and vecuronium) at various doses in adults who are undergoing general elective surgery with sevoflurane anesthesia.

Study participants received an intubating dose of a neuromuscular blocker (to enable insertion of a tube through the nose or mouth into the trachea to provide artificial ventilation). The intubating dose was followed by repeated bolus maintenance doses as needed, to maintain muscle relaxation. The time it takes to reach maximal effect of the neuromuscular blocker (onset time) after the intubating dose was measured and compared as the primary outcome.

DETAILED DESCRIPTION:
The TOF Watch-SX (acceleration transducer) was used in the measurement of neuromuscular blocking action.

ELIGIBILITY:
Inclusion criteria:

* at least 20 but under 65 years of age
* American Society of Anesthesiologists (ASA) Class 1, 2 or 3 for general elective surgery
* not considered to be pregnant
* scheduled for elective surgery under sevoflurane or propofol anesthesia with an anticipated duration of about 1.5-3 hours
* normal laboratory values

Exclusion Criteria:

* certain medical conditions or medical histories
* receiving certain medications or treatments

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2003-02; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Onset time of intubating dose. DESCRIPTION: The time interval between the completion of injection of the study drug (rocuronium or vecuronium) and the maximal depression of first twitch--measured via TOF Watch Sx(R)-- was defined as the onset time. | Day of Surgery, after injection of study drug until maximal depression of first twitch achieved

SECONDARY OUTCOMES:
Number of subjects who achieved maximal block >=90% after the intubating dose. DESCRIPTION: Reaching a 90% depression of first twitch--measured via TOF Watch Sx(R)--was defined as achieving 90% block | Day of Surgery, after injection of study drug until maximal depression of first twice achieved
Clinical duration after first maintenance dose. DESCRIPTION: The time interval between the completion of injection of study drug and return of first twitch to 25%(as measured by TOF Watch Sx(R)) was defined as the clinical duration. | Day of Surgery, after injection of study drug until return of first twitch to 25%